CLINICAL TRIAL: NCT00238810
Title: Retrospective Evaluation of Serum B-type Natriuretic Peptide Hormone Levels in Post-operative Patients and the Relationship of BNP Levels to Cardiac Diagnosis, Operation Performed, Post-operative Course and Outcome
Brief Title: Relationship of Brain Natriuretic Peptide (BNP) Levels to Cardiac Diagnosis, Operation Performed, Post-operative Course and Outcome
Status: Completed | Type: Observational
Sponsor: Children's Healthcare of Atlanta (Other)
Responsible Party: Sponsor
Other Study IDs: 05.068
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Heart Disease
Keywords: BNP; Pediatrics; Congenital heart disease; b-type natriuretic peptide
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to assess brain natriuretic peptide levels to evaluate the relationship of those levels with the diagnosis of congenital cardiac disease, operation performed, post-operative course, and outcome.

DETAILED DESCRIPTION:
Three types of natriuretic peptides (NP) have been isolated: atrial natriuretic peptide (ANP), brain natriuretic peptide (BNP), and C-type natriuretic peptide (CNP). The NP family elicits a number of vascular, renal and endocrine effects that help to maintain blood pressure and extracellular fluid volume. These effects are mediated by the specific binding of NP to cell surface receptors that have been characterized, purified and cloned from cells of the vasculature, kidney, adrenal gland and brain. There are 3 subtypes of NP receptors: type A natriuretic peptide receptor (NPRA), type B natriuretic peptide receptor (NPRB), and type C natriuretic peptide receptor (NPRC). All 3 subtypes affect cellular second messenger activity. The literature currently does not define the levels of b-type natriuretic peptide (BNP) in children with congenital heart disease undergoing surgery.

The investigator wishes to perform a retrospective chart review to define BNP levels in the pediatric cardiac defect population and to evaluate the relationship of those levels with cardiac diagnosis, operation performed, post-operative course and outcome. The investigator will collect the following information from the medical record:

* Laboratory: BNP levels, serum pH, lactic acid, Co-ox, CBC, Chemistry
* Diagnosis
* Surgical Procedure
* Incidence of re-operation
* Length of ICU Stay
* Length of Hospital Stay
* Complications
* Length of Ventilation (how many days on the ventilator)
* Medications
* Cross Clamp Time
* Bypass Time
* Echocardiogram data
* Cardiac Catheterization Data
* Vital Signs
* Monitored Hemodynamic Measures
* Final outcome (discharged or death)

ELIGIBILITY:
Inclusion Criteria:

* Congenital heart defect

Exclusion Criteria:

* Patients without congenital heart defects

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with congenital heart defects
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2005-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
define BNP levels in the pediatric cardiac defect population and to evaluate the relationship of those levels with cardiac diagnosis, operation performed, post-operative course and outcome. | 9 years
  define BNP levels in the pediatric cardiac defect population and to evaluate the relationship of those levels with cardiac diagnosis, operation performed, post-operative course and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alecia Wang, MD, Principal Investigator — Emory University Cardiac Fellow at Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Nakayama T. The genetic contribution of the natriuretic peptide system to cardiovascular diseases. Endocr J. 2005 Feb;52(1):11-21. doi: 10.1507/endocrj.52.11. PMID 15758553